CLINICAL TRIAL: NCT06097507
Title: Patient and Prescriber Perspective on Climate Impact of Inhalers in the Treatment of Asthma
Brief Title: Patient Perspective on Climate Impact of Inhalers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nicole Ezer, MD, FRCPC, MPH, MDCM, FRCPC, MPH, Assistant professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-10072
Record Dates: First submitted 2023-10-11; First posted 2023-10-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: Asthma; Inhalers; Environment; Climate impact
MeSH Terms: conditions — Asthma | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Asthma patients (Experimental): Low risk educational intervention. The consented patients will be given an information packet containing an infographic about the climate impact of inhalers, a letter explaining the option of changing inhalers (which clearly outlines that the Bricanyl Turbuhaler will not cost them more money than the Ventolin) and a pre-filled prescription for Bricanyl Turbuhaler.
  Also 5 selected asthma providers will be asked to fill a questionnaire on their perspectives on the climate impact of inhalers and their approach to inhaler rotation. This may also be supplemented with a phone interview
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — The consented patients will be given an information packet containing an infographic about the climate impact of inhalers, a letter explaining the option of changing inhalers (which clearly outlines that the Bricanyl Turbuhaler will not cost them more money than the Ventolin) and a pre-filled prescription for Bricanyl Turbuhaler.

SUMMARY:
The effects of climate change on population health have considerably increased as the planet warms and is thus subjected to more heat waves, extreme weather events and food insecurity. Paradoxically, healthcare systems are major contributors to carbon emissions.

Within the field of respirology, choice of inhaler is a low-hanging fruit to address this issue. Metered dose inhalers (MDI) contain potent greenhouse gases and have been shown to have a significantly larger carbon footprint than dry powder inhalers (DPI).

The goal of the study is to assess asthma patients' willingness to change inhalers for environmental reasons as well as prescribers' willingness to prescribe a different inhaler for environmental reasons at the patient's request. The study will also be assessing patient awareness of the climate impact of inhalers and the importance that they attribute to this issue as well as other issues (cost and ease of use).

DETAILED DESCRIPTION:
The effects of climate change on population health have considerably increased as the planet warms and is thus subjected to more heat waves, extreme weather events and food insecurity. Paradoxically, healthcare systems are major contributors to carbon emissions.

Within the field of respirology, choice of inhaler is a low-hanging fruit to address this issue. Metered dose inhalers (MDI) contain potent greenhouse gases and have been shown to have a significantly larger carbon footprint than dry powder inhalers (DPI).

Studies from the United Kingdom have revealed that although patient awareness of the discrepancy in climate impact of inhalers is low, their willingness to change inhalers after being educated on the subject is high.

An example of inhaler change is to use the Bricanyl Turbuhaler (terbutaline) instead of Ventolin (salbutamol) as a rescue medication in asthma. They are both short-acting bronchodilators (SABA) and have similar pharmacodynamics. However, use of Bricanyl for one year produces 7,183 kgCO2e or the equivalent of 59.9km by car, whereas use of Ventolin for one year produces 411,720 kgCO2e, the equivalent of 3,431 km by car.

The goal of the study is to assess asthma patients' willingness to change inhalers for environmental reasons as well as prescribers' willingness to prescribe a different inhaler for environmental reasons at the patient's request. The study will also be assessing patient awareness of the climate impact of inhalers and the importance that they attribute to this issue as well as other issues (cost and ease of use).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Followed in the asthma clinic at the Montreal Chest Institute or the Montreal General Hospital.
* Confirmed diagnosis of asthma presenting for a follow up visit for their asthma (defined as positive methacholine challenge test or confirmed reversibility of lung function 12% increase FEV1 (forced expiratory volume) or 200ml absolute value increase post bronchodilator).
* On an inhaled steroid for the treatment of asthma for maintenance as well as Ventolin MDI as a rescue inhaler.
* Stable asthma -not currently being evaluated for an acute asthma exacerbation and no Emergency Room visits for asthma within the last 30 days.
* Adequate lung function with a FEV1 of at least 50% and, where available, a peak inspiratory flow (PIF) of under 60L/m for use of a DPI and MDI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Rotation of Ventolin MDI to Bricanyl Turbuhaler. | 30 days
  Proportion of participants who changed their inhaler from Ventolin MDI to Bricanyl Turbuhaler within 30 days of study visit.

SECONDARY OUTCOMES:
Rate of failure of the intervention | 90 days
  defined as a rotation back from Bricanyl to Ventolin MDI within 90 days after the clinic
Proportion of patients who filled Bricanyl Rx change | 30 days
  Proportion of patients who filled Bricanyl Rx change with pharmacist within 30 days of the clinic but did not possess the medication (30 day medication possession ratio)
Awareness of patients regarding the climate impact of inhalers | Baseline
  Awareness of patients regarding the climate impact of inhalers defined by questionnaire data, using a 5 point likert scale (from "not at all aware" to "extremely aware")
Patients' willingness to change inhalers for environmental reasons | Baseline
  Patients' willingness to change inhalers for environmental reasons and the importance of different issues (environmental impact, cost, ease of use) for patients, using 3 different 5 point likert scale, one for each sub-category)
Providers' willingness to change inhalers for environmental reasons | 6 months
  Providers' willingness to change inhalers for environmental reasons and the importance of different issues (environmental impact, cost, ease of use) for patients.
  This will be assessed through 5 different 5 points likert scale, as well as with a phone interview.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No